CLINICAL TRIAL: NCT05560828
Title: A Multi-centre Cohort Study Comparing Health Outcome Data From Holter Monitoring to 14 Day Zio Monitoring in People Where Ambulatory ECG Monitoring is Required
Brief Title: Zio Real-World Evaluation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: KCLAI001
Record Dates: First submitted 2022-08-16; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Cardiology; Stroke/TIA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zio Cohort: Patients who have been prescribed Zio
  Interventions: Other: Zio XT service
- Holter Cohort: Patients who have been prescribed Holter

INTERVENTIONS:
Other: Zio XT service — There will be no intervention. Standard of care at participating NHS organizations will not be affected.
  Groups: Zio Cohort

SUMMARY:
In 2020 an independent evaluation of the Zio service as part of the Digital Health Technologies programme at NICE was conducted. From the available clinical and economic evidence, the evaluation concluded that further evidence is needed to estimate the resource use associated with Zio compared with standard care, particularly the number of outpatient visits and repeat testing needed. Additionally it recommended further evidence is needed for the longer-term clinical consequences such as anticoagulant uptake and other changes to treatment related to the results from monitoring. (MTG52) Therefore, this study aims to address these uncertainties and identify whether the Zio service could be used in the health and social care system in England. This will be assessed using a multicentre, cohort study design consisting of two cohorts. The data for the existing standard of care cohort using Holter monitor (cohort 1) will be collected from 6-month retrospective pre-covid data, and, for the Zio service cohort (cohort 2), data will be collected retrospectively over a 6-month period. Each cohort will include two separate populations recruited from cardiology clinics and stroke/TIA clinics. The main objective of this study is to analyse quantitative data collected from participating sites and complementary qualitative data on Zio utilisation from questionnaires

DETAILED DESCRIPTION:
The proposed study is a multi-centre, cohort study that will collect 6-month control data from a cohort of participants wearing Holter devices (2018-2019) and match this data to a 6-month cohort of patients wearing Zio patches (2021 - 2022). An additional cohort of patients using the Zio patch from both the cardiology and stroke/TIA population will be included for the patient experience aspect of the study.

Other designs have been considered but from a pragmatic point of view and the need for a "real-world" evaluation this is the preferred alternative with the caveat that there may not be an exact match between the two patient groups.

The proposed study is a multi-centre, cohort study that will collect 6-month baseline data from a retrospective cohort of participants wearing Holter devices and match this data to a 6-month retrospective cohort of patients wearing Zio patches. Zio is standard of care at the NHS sites participating in this study, but it is not standard of care across the NHS. The standard of care received by patients involved in this study will not be affected by their participation in the study. However, should Zio be adopted more widely by the NHS, a change in pathway will be required. The Zio device is CE marked as a Class IIa and will be used within its intended purpose.

Two separate populations will be considered for this study: cardiology outpatients and patients at risk of (or who have had a previous) stroke or TIA. Each of these populations will comprise a control cohort for Holter monitor and a cohort for Zio service, which will be analysed separately. A separate cohort comprising of participants prescribed Zio will be included in a qualitative analysis to assess their experience of using Zio and previous experience of using Holter monitor within the past 2 years, where applicable. This will allow for a comparative analysis of patient experience. For patients in the cohort who have not had prior experience of using Holter monitor, a questionnaire will be administered to assess their experience of using Zio only.

Given the potential for a shift in the spectrum of the population that may be expected when Zio is implemented, propensity score matching will be utilised to compare the Holter and Zio cohorts for both the stroke/TIA and cardiology arms.

ELIGIBILITY:
Inclusion Criteria:

Data from stroke/TIA population:

* 18 years of age or older
* diagnosed with having had an ischaemic non-lacunar stroke or probable TIA by a stroke clinician or neurologist.
* Referred for ambulatory ECG monitoring

Data from cardiology population:

* 18 years of age or older
* experiencing symptomatic palpitations, dizziness, pre-syncope or syncope
* Referred for ambulatory ECG monitoring

Qualitative data will be collected via self-administered questionnaires from healthcare professionals who:

• are involved in prescribing the Zio XT service, fitting the Zio patch, interpreting the Zio report and making a treatment decision.

Qualitative data will be collected via self-administered questionnaires from patients who:

* are 18 years of age or older
* have been prescribed the Zio patch
* have been prescribed the Zio patch and the Holter monitor (within two years)

Exclusion Criteria:

Data from stroke/TIA population:

* History of AF or atrial flutter
* > 50% stenosis of a potentially symptomatic cervical artery (carotid or vertebral)
* Pre-existing indication or contraindication for permanent anticoagulation therapy
* Significant uncertainty of TIA diagnosis such as cases where TIA treatment isn't initiated
* New lacunar stroke reported on imaging which corresponds to the presenting stroke syndrome

Data from cardiology population:

* Patients in whom 24-hour monitoring is required due to the following reasons:

  * experiencing daily symptoms
  * the need for AF rate control measurement
  * the need for ectopic burden measurement
* Patients who are prescribed Implantable Loop Recorders and pacemakers in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two cohorts will be recruited from a cardiology and stroke/TIA population
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to device being fitted | 6 months
  Time to device being fitted
Time to diagnosis | 6 months
  Time to diagnosis
Time to treatment decision | 6 months
  Time to treatment decision - referral for anticoagulant prescription or other clinical intervention, where needed

SECONDARY OUTCOMES:
Resource utilisation | 6 months
  Resource utilisation
Time to ECG report | 6 months
  Time to ECG report
Time to repeat ambulatory ECG test referrals | 6 months
  Time to repeat ambulatory ECG test referrals
Number of insertable cardiac monitors such as LINQ implants | 6 months
  Number of insertable cardiac monitors such as LINQ implants
Number of hospital visits | 6 months
  Number of hospital visits
Number of inconclusive follow-up appointments | 6 months
  Number of inconclusive follow-up appointments
Number of device failures / adverse events | 6 months
  Number of device failures / adverse events
Proportion of patients that undergo full monitoring following referral | 6 months
  Proportion of patients that undergo full monitoring following referral
Diagnostic yield | 6 months
  Diagnostic yield
"Rule out" | 6 months
  "Rule out" - number of patients with non-clinically significant arrhythmia
Time to discharge of patients with non-clinically significant cardiac arrhythmia | 6 months
  Time to discharge of patients with non-clinically significant cardiac arrhythmia
Settlement of patient's GP surgery - urban or rural area | 6 months
  Settlement of patient's GP surgery - urban or rural area
Patient experience | 6 months
  Patient experience of using Zio
Clinical experience of using Zio | 6 months
  Clinical experience of using Zio

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared